CLINICAL TRIAL: NCT01416987
Title: A Korean Post-Marketing Surveillance Study On Pergoveris® (Follitropin Alfa + Lutropin Alfa)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200061-507
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — pergoveris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Pergoveris® — Participants received once daily injection of a single vial of Pergoveris® which contained 150 International Units (IU) of follitropin alfa (r-hFSH) and 75 IU of lutropin alfa (r-hLH), for approximately 8 days.

SUMMARY:
This prospective study collected safety information from more than 600 participants treated with Pergoveris®.

During the Post-Marketing Surveillance (PMS) period, data about the participant's background, participant's medical history, Pergoveris® indication, prior infertility medication, Pergoveris® treatment status, concomitant drugs, all adverse events (regardless of the causal relationship to Pergoveris®) and efficacy (follicular growth and clinical pregnancy) were collected for study purposes.The post marketing surveillance was based on all cases treated with Pergoveris®.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who were eligible for Pergoveris® treatment according to the indication in the national label of Pergoveris®. The national label approved by Korea Food & Drug Administration is "Pergoveris® in association with a follicle stimulating hormone(FSH) preparation was recommended for the stimulation of follicular development in women with severe Luteinizing Hormone (LH) and FSH deficiency. In clinical trials these participants were defined by an endogenous serum LH level less than (<)1.2 International units per liter IU/L"

Exclusion Criteria:

* According to national label

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertile participants
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-08-14 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd.
Locations (1):
- Research site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pergoveris®
Started | 600
Completed | 600
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of Pergoveris®.
Arm/Group | Pergoveris®
Number analyzed (Participants) | 600
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.58 (3.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 600
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event (AE) and Adverse Drug Reaction (ADR)
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Adverse events included both Serious AEs and non-serious AEs. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Adverse Drug Reactions (ADR) was defined as an adverse event for which a causal relationship between the product and the occurrence was suspected, that was judged possible or probable by the reporting physician.
Time Frame: 2463 days
Population: Safety analysis set included all participants who received at least one dose of Pergoveris®.
Measure: Count of Participants; unit: Participants
Arm/Group | Pergoveris®
Number analyzed (Participants) | 600
Participants
  Adverse event (AE) | 16
  Adverse drug reaction (ADR) | 13

2. Secondary Outcome: Number of Participants With at Least One Follicle of More Than 17 Millimeter (mm) of Mean Diameter on Ultrasonography
Description: Number of participants with one follicle of more than 17mm of mean diameter on ultrasonography were reported.
Time Frame: 2463 days
Population: Effectiveness analysis set included participants who were evaluated for follicular growth (FG) after treatment with Pergoveris®, except those; who were not assessed for FG; whose assessments of FG were considered 'undecidable' based on Human Chorionic Gonadotropin (HCG) not administered, ultrasonography not done on the day of HCG administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Pergoveris®
Number analyzed (Participants) | 532
Participants | 528

3. Secondary Outcome: Number of Participants With Clinical Pregnancy as Per Safety Analysis Set
Description: The clinical pregnancy was defined as a positive serum in urine HCG test or as the presence of gestational sac or yolk sac by an ultrasonography confirmation.
Time Frame: 2463 days
Population: Safety analysis set included all participants who received at least one dose of Pergoveris®.
Measure: Count of Participants; unit: Participants
Arm/Group | Pergoveris®
Number analyzed (Participants) | 600
Participants | 246

4. Secondary Outcome: Number of Participants With Clinical Pregnancy as Per Effectiveness Analysis Set
Description: as for outcome 3
Time Frame: 2463 days
Population: Effectiveness analysis set included participants who were evaluated for follicular growth (FG) after treatment with Pergoveris ®, except those; who were not assessed for FG; whose assessments of FG were considered 'undecidable' based on Human Chorionic Gonadotropin (HCG) not administered, ultrasonography not done on the day of HCG administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Pergoveris®
Number analyzed (Participants) | 532
Participants | 227

ADVERSE EVENTS:
Time Frame: 2463 days
Arm/Group | Pergoveris®
All-Cause Mortality (participants affected / at risk) | 0/600
Serious Adverse Events (participants affected / at risk) | 2/600
Other Adverse Events (participants affected / at risk) | 14/600
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pergoveris® (N=600)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pergoveris® (N=600)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Injection site erythema (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site pruritus (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT01416987/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT01416987/SAP_001.pdf